CLINICAL TRIAL: NCT07362147
Title: Exploring the Effects of Hand and Foot Exercise Intervention in Older Adults With Gynecological Cancer Receiving Chemotherapy Improvement of Peripheral Neuropathy and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-12-008A
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Neuropathy; Cervical Cancer; Endometrial Cancer; Ovarian Cancer; Vaginal Cancers; Fallopian Tube Cancers
Keywords: hand and foot exercises, chemotherapy, gynecological cancer, peripheral neuropathy, quality of life
MeSH Terms: conditions — Peripheral Nervous System Diseases; Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Intervention Model Description: The experimental group received 12 weeks of hand and foot movement interventions (10-15 min/session * 3 sessions/week).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- experimental group (Experimental)
  Interventions: Other: hand and foot exercises

INTERVENTIONS:
Other: hand and foot exercises — The hand and foot exercise steps include hand and foot movements, practiced in a seated position. Hold each movement for ten seconds and then relax, repeating ten times. Perform the hand and foot exercises three times a day, for 10-15 minutes each time, three days a week, for twelve weeks.
  Arms: experimental group

SUMMARY:
Paclitaxel-based drugs are commonly used adjuvant chemotherapy for gynecological cancer patients. Peripheral neuropathy, a side effect of this treatment, presents with symptoms such as numbness, tingling, decreased skin and reflex sensation, and impaired function in the hands and feet, thus affecting quality of life. Peripheral neuropathy is a side effect caused by the neurotoxicity of certain chemotherapeutic drugs, including paclitaxel and platinum-based drugs, resulting from the cumulative toxicity of specific drug doses. While numerous international studies have confirmed the preventative effects of hand and foot movement interventions, there is a lack of relevant literature in China. Therefore, this study aims to explore the effects of hand and foot movement interventions on elderly gynecological cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Peripheral neuropathy is a fairly common clinical problem. Paclitaxel-based drugs are commonly used adjuvant chemotherapy for gynecological cancer patients, and peripheral neuropathy symptoms, including numbness, tingling, decreased skin and reflex sensation, and impaired function, can significantly impact quality of life. Peripheral neuropathy is a side effect caused by the neurotoxicity of certain chemotherapeutic drugs, including paclitaxel (Paclitaxel, Docetaxel) and platinum-based drugs (Cisplatin, Carboplatin). It results from the cumulative toxicity of specific drug doses. A study by Eroglu & Kutluturkan (2024) showed that in colorectal cancer patients receiving at least two cycles of platinum-based drugs, a hand and foot exercise program performed three times daily, three days a week, for eight weeks effectively reduced sensory and motor symptoms of peripheral neuropathy, as well as the severity, frequency, and emotional distress caused by symptoms, and the impact of symptoms on hand and foot dexterity. Another study reported that breast cancer patients receiving paclitaxel chemotherapy and diagnosed with grade I or higher neuropathy benefited from massage or stress ball exercises for eight weeks. These exercises helped reduce the incidence and severity of peripheral neuropathy during and after chemotherapy, prevented muscle weakness caused by peripheral neuropathy, and improved independent function and quality of life (Uysal & Toprak, 2025). Currently, there is a lack of empirical research in China on using hand-foot exercise interventions to improve peripheral neuropathy and quality of life in gynecological cancer patients undergoing chemotherapy, and care guidelines are severely lacking. More research is needed to confirm its efficacy. Therefore, this study aims to explore the effectiveness of hand-foot exercise interventions in improving peripheral neuropathy and quality of life in elderly gynecological cancer patients undergoing chemotherapy. Currently, many studies abroad have confirmed that hand and foot exercise intervention can effectively prevent [the condition]. We would like to invite you to participate in a research trial. You are free to decide whether or not to participate in this trial. Before receiving the hand and foot exercise at our hospital's obstetrics and gynecology outpatient clinic, we will explain the process and obtain your consent. We will provide you with a paper picture booklet of hand and foot exercises. After the researcher demonstrates the hand and foot exercise instructions to the participant using a massage ball, the researcher and the participant will perform the hand and foot exercises together one-on-one to confirm that the participant's movements are performed correctly. You can also watch the hand and foot exercise instructional video online. At the same time, you will be given a weekly exercise record sheet, indicating whether you have completed the exercise by checking a box. Participants will then perform the hand and foot exercises at home for 10-15 minutes each time, three times a day, three days a week, for twelve weeks. After that, you will return the exercise record sheet.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 65 or older diagnosed with gynecological cancer (stage II to IV) by a physician, without skin or nail lesions.

Individuals who have received at least one course of chemotherapy within the past year and have peripheral neuropathy, with chemotherapy drugs including paclitaxel (Paclitaxel or Docetaxel) or platinum-based drugs (Cisplatin or Carboplatin), and may receive combined targeted or immunotherapy.

Individuals who are conscious and able to communicate in Mandarin, Taiwanese, or written language.

Exclusion Criteria:

Skin or nail lesions. Edema of 3+ or more in the extremities. History of diagnosis of diabetes, neuropathy, peripheral arterial ischemia, or multiple organ failure.

Distal bone or skin metastases. Patients who have interrupted chemotherapy. Patients who have participated in similar studies.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral neuropathy | From enrollment to the end of treatment at 12 weeks.
  The content includes FACT/GOG-Ntx variable data.The maximum score is 120 points, and the minimum score is 0 points.A higher score indicates a better result.

SECONDARY OUTCOMES:
Quality of life | From enrollment to end of treatment (12 weeks)
  The content includes EORTC QLQ-CIPN20 variable data.The maximum score is 100 points, and the minimum score is 0 points. A higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: CHANG Chen Hsuan, Study Chair
Locations (1):
- Taipei Veterans General Hospital, Taipei, No.201, Sec. 2, Shipai Rd., Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eroglu I, Kutluturkan S. The effect of hand-foot exercises on chemotherapy-induced peripheral neuropathy-related pain, falls, and quality of life in colorectal cancer: A randomized controlled trial. Eur J Oncol Nurs. 2024 Aug;71:102641. doi: 10.1016/j.ejon.2024.102641. Epub 2024 Jun 15. PMID 38897103
- See also: This study followed the hand and foot movement guidelines recommended by Eroglu & Kutluturkan (2024). Because the guidelines are relevant to the specific conditions of the cases in this study. — https://drive.google.com/file/d/1H7B3UzqRn8WV4pzZZQ0U-G4KFyoOXlFn/view